CLINICAL TRIAL: NCT03257527
Title: Enduring Happiness and Continued Self-Enhancement (ENHANCE) 2.0: A Well-Being Program
Brief Title: Enduring Happiness and Continued Self-Enhancement (ENHANCE) 2.0
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Frank C. Diener Foundation (Unknown); University of Virginia (Other); University of Utah (Other)
Responsible Party: Principal Investigator, Lesley Lutes, Associate Professor, Director of Clinical Training, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H16-02273
Record Dates: First submitted 2017-08-08; First posted 2017-08-22 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Well-being
Keywords: Well-being; Comparative Clinical Trial; Positive Psychology Intervention; Mindfulness Based Stress Reduction (MBSR); Group Therapy; Happiness; Bibliotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ENHANCE group (Experimental): The ENHANCE group is comprised of 12 weekly session to be completed in-person and delivered by trained group facilitators.
  Interventions: Behavioral: ENHANCE group
- MBSR group (Active Comparator): The MBSR group will complete a self-help workbook entitled, "A Mindfulness-Based Stress Reduction Workbook" over a 12 week period.
  Interventions: Behavioral: MBSR group

INTERVENTIONS:
Behavioral: ENHANCE group — The ENHANCE program includes an initial 3-month treatment of 12 weekly sessions (including an introductory session, a final session, and 10 content sessions) followed by a 3-month maintenance phase intervention with bi-weekly sessions. Over the course of the program, participants will learn about 10 evidenced-based principles of happiness and how these principles can be applied effectively in their lives. At the final session, participants will receive feedback outlining the happiness principles and activities that fit them best, and will then be asked to work on creating a plan for integrating those principles into their daily lives.
  Arms: ENHANCE group
Behavioral: MBSR group — The MBSR program is based on the self-help workbook entitled, "A Mindfulness-Based Stress Reduction Workbook". This workbook is authored by Drs. Bob Stahl and Elisha Goldstein - who are both certified MBSR trainers. The workbook is written to help everyday people learn how to replace stress-promoting habits with mindfully-based ones to improve overall well-being. The workbook begins by providing a thorough introduction to the basic tenets of mindfulness, and improving well-being through the use of mindfulness-based skills. The workbook outlines, in detail, several skills-based exercises for practicing mindfulness across different aspects of a person's life. The MBSR group will be provided with a recommended weekly schedule for the initial 3-month treatment and a list of additional resources to be completed over the 3-month maintenance phase.
  Arms: MBSR group

SUMMARY:
The study is designed to compare the efficacy of two programs intended to improve happiness and well-being among healthy, community adults between the ages of 25 and 75 years. Participants will complete either an in-person program (ENHANCE) or a mindfulness-based stress reduction (MBSR) self-help program over 3-months. The ENHANCE program will include 12-weekly sessions based on researched principles of happiness. Alternatively, the MBSR self-help guide will teach ways to replace stress-promoting habits. Participants will be asked to complete a series of measures at three points of the study: at the start of the study, the end of the study, and 3-months following the study.

DETAILED DESCRIPTION:
In 2011, the United Nations defined happiness as a "fundamental human goal" and invited Member States to pursue measures that enhance the happiness of their citizens. The majority of people across the globe agree that happiness is an important goal. In accordance with this global goal to be happy, the psychological literature abounds with interventions to combat problems that may prevent people from being happy-from obesity to depression and physical pain. However, happiness is not simply the absence of problems. Yet, interventions to help people attain and maintain higher levels of happiness are rare. Accordingly, in a previous study, the investigators designed and evaluated the efficacy of a theoretically-grounded, evidence-based randomized controlled trial for enhancing happiness and well-being. In the present study, it is the goal to assess the efficacy of modifications made to the original program, and compare the program to a self-help comparison group. All participants in the study will complete weekly questionnaires, as well as the same battery of online assessments at baseline, the end of the study, and 3-months following the study. The investigators will be examining if changes seen from baseline to the end of the interventions are maintained through a maintenance intervention in both arms for 3 months following the primary intervention.

It is expect that participants actively completing the in-person ENHANCE program will report greater increase in their overall levels of happiness/well-being at the end of the 12-week program compared to participants in the MBSR self-help group. It is predicted that there will be a downstream effect on happiness for all participants' mental and physical health, cognitive function, social relationships, and other positive outcomes, but that this effect will be greater for participants in the active in-person ENHANCE group. The insights gained from this research could be used in future intervention research towards promoting health, achievement, citizenship, and better relationships.

ELIGIBILITY:
Inclusion Criteria:

* All participants in the study will include males and females between the ages of 25 and 75 years. Participants of all racial and ethnic backgrounds will be eligible to participate. Participants of all religious and spiritual orientations will be eligible to participate.

Exclusion Criteria:

* Participants will be screened for major psychological disorders, such as anxiety and depression using the Patient Health Questionnaire-9 (PHQ-9. Participants who are screened with a major mental illness (such as severe depression as determined by a cut-off score of 15 or greater on the PHQ-9) will be advised that this study is not designed as a treatment for mental illness (including severe depression), and will be given a list of the appropriate mental health services offered in their community (e.g., Kelowna Mental Health and Substance Use Services).

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Satisfaction With Life | Baseline, 3, 6 months
  Satisfaction With Life Scale
Change from Baseline in Positive Affect | Baseline, 3, 6 months
  Scale of Positive and Negative Experience: SPANE
Change from Baseline in Negative Affect | Baseline, 3, 6 months
  Scale of Positive and Negative Experience: SPANE
Change from Baseline in Meaning in Life | Baseline, 3, 6 months
  Meaning in Life Questionnaire
Change from Baseline in Thriving | Baseline, 3, 6 months
  Comprehensive Inventory of Thriving

SECONDARY OUTCOMES:
Change from Baseline in Physical Activity | Baseline, 3, 6 months
  Step count captured from Fitbits
Change from Baseline in Perceived Social Support | Baseline, 3, 6 months
  The Social Provisions Scale
Change from Baseline in Relationship Satisfaction | Baseline, 3, 6 months
  The Revised Dyadic Adjustment Scale
Change from Baseline to attention, concentration, reaction time, memory, processing speed, executive functioning and decision-making | Baseline, 3, 6 months
  Automated Neuropsychological Assessment Metrics (ANAM)
Change from Baseline in Implicit Theories of Well-Being | Baseline, 3, 6 months
Change from baseline to Empathy | Baseline, 3, 6 months
  The Toronto Empathy Questionnaire

OTHER OUTCOMES:
Change from Baseline Positive and Negative Memories Generated by Participants | Baseline, 3, 6 months
  In this task, participants list as many positive (and then negative) life events and then as many negative life events as they can in three minutes. Relative quantities of positive to negative life events that are listed demonstrate accessibility of positive and negative memories, which is an indicator of Subjective Well-Being.
Change from Baseline Peer Reports of Positive Behaviors | Baseline, 3, 6 months
  Peers will be asked to evaluate the participant on how frequently they engaged in a series of affect-related displays over the past week: smiling, laughing
Change from Baseline Peer Reports of Satisfaction With Life | Baseline, 3, 6 months
  Peers will be asked to report on changes to the participant's satisfaction with life
Change from Baseline Peer Reports of Positive Affect | Baseline, 3, 6 months
  Peers will be asked to report on changes to the participant's positive affect
Change from Baseline Peer Reports of Negative Affect | Baseline, 3, 6 months
  Peers will be asked to report on changes to the participant's negative affect
Change from Baseline Peer Reports of Negative Behaviors | Baseline, 3, 6 months
  Peers will be asked to evaluate the participant on how frequently they engaged in a series of affect-related displays over the past week: crying, frowning, complaining, and criticizing
Change from Baseline Healthy Behaviors | Baseline, 3, 6 months
  Behavioral Risk Factor Surveillance System
Change from Baseline Perceived Stress | Baseline, 3, 6 months
  Perceived Stress Scale (PSS)
Change from Baseline Depression | Baseline, 3, 6 months
  Patient Health Questionnaire-9
Change from Baseline Self-Esteem | Baseline, 3, 6 months
  Rosenberg Self-Esteem Scale
Change from Baseline Psychological Need Satisfaction: Autonomy, Competence, Relatedness | Baseline, 3, 6 months
  Need Satisfaction Scale
Change from Baseline Body Mass Index: BMI | Baseline, 3, 6 months
  BMI = (Weight in Kilograms / (Height in Meters x Height in Meters))
Change from Baseline Blood Pressure | Baseline, 3, 6 months
  Blood pressure is taken twice using a blood pressure cuff and the average will be reported
Change from Baseline Sleep Quality | Baseline, 3, 6 months
  The Pittsburgh Sleep Quality Index
Change from Baseline Alertness | Baseline, 3, 6 months
  The Stanford Sleepiness Scale
Objective Change from Baseline in Sleep | Baseline, 3, 6 months
  Fitbit Sleep data: length, # of times awake

CONTACTS AND LOCATIONS:
Locations (1):
- University of British Columbia Okanagan, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided
We are currently consulting with others on the grant team regarding our long-term data plan and will update with our final data sharing plan in October 2017